CLINICAL TRIAL: NCT03464214
Title: The Effects of Local Vibration and Cervical Stabilization Exercises Applied on Neck Muscles on Balance in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Turkmen, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 15/716-04
Record Dates: First submitted 2018-02-27; First posted 2018-03-13 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cervical Pain; Somatosensory Disorders; Vestibular Diseases
Keywords: Vibration; Cervical stabilization exercises; Physiotherapy and rehabilitation; Sensory organization test; Balance
MeSH Terms: conditions — Neck Pain; Somatosensory Disorders; Vestibular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibration Group (Active Comparator): Local vibration on neck muscles
  Interventions: Device: Neck Muscle Vibration
- Stabilization Group (Active Comparator): Cervical stabilization exercises on cervical region
  Interventions: Behavioral: Cervical Stabilization Exercises
- Control Group (No Intervention): Individuals performed only daily living activities

INTERVENTIONS:
Device: Neck Muscle Vibration — Local vibration device applied on neck muscles for 8 weeks
  Arms: Vibration Group
Behavioral: Cervical Stabilization Exercises — Cervical stabilization exercises performed by healty individuals for 8 weeks
  Arms: Stabilization Group

SUMMARY:
In healthy individuals, many postural musculoskeletal problems arise due to various reasons. The cervical region is the region where these problems are most common. The cervical region ranks second in the general population after the lumbal area of musculoskeletal system disorders and affects close to 70% of the general population.The most important causes of this posture disorder are; muscular performance and strength are inadequate, as well as decreased proprioception of the muscles, deterioration of the individual balance systems that result in individual visual or vestibular problems.

Exercise therapy is at the forefront of these methods, while a variety of methods are applied in the prevention and treatment of neck problems. Recent studies have focused on multifaceted treatments including exercises to improve strength, endurance and coordination of cervical muscles, proprioceptive training, relaxation exercises to prevent muscle tension, stabilization exercises and behavior modification. Cervical stabilization exercises are a frequently used exercise approach. Cervical stabilization exercises, which are different from ordinary exercises, are based on biomechanics, neurophysiology and physiotherapy research. The main objective of this method is; improve body awareness, maintain posture uniformity, improve strength, endurance, coordination and proprioception. Stabilization exercises also increase the strength and endurance of the postural and stabilizer muscles, improving stability control in the stabilized and non-stabilized positions.

Another method that contributes to the development of balance and proprioceptive sense is vibration application. Proprioception plays an important role in ensuring the coordination of movements. When the proprioception input is disturbed, both the position sense and the speed of movement may be affected. Muscle-tendon vibration is a noninvasive method that is often used in proprioception studies. It has been suggested that the vibration application are the enhancing effect of the proprioceptive. However, there is not enough research on this subject.

The purpose of this study is to determine whether the cervical stabilization exercises to be applied to the cervical region and the local vibration applied to the neck muscles are related to muscle performance, proprioception and balance and their superiority with each other.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have not had neck pain in the last six months.

Exclusion Criteria:

* Patients with atypical spinal cord anomalies, inflammatory or rheumatologic disorders, malignancy history, radiculopathy, myelopathy or other neurological disorders, vestibular disorders, and vertebral trauma history who underwent any surgical treatment for vertebral colonic at least 3 months before, was not included in the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03-12 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Sensory Organization Test | SOT was used to assess changes in visual, vestibular, and somatosensory balance of individuals at eighth week.
  The sensory organization test. The sensory organization test (SOT) was developed to describe the contribution levels of the three basic systems of balance (visual, vestibular, somatosensory) to the general equilibrium. SOT was used to assess changes in visual, vestibular, and somatosensory balance of individuals at eighth week.

SECONDARY OUTCOMES:
Head Shake Sensory Organization Test (HS-SOT) | HS-SOT was used to assess changes only vestibular balance of individuals at eighth week.
  This test is applied in the second and fifth cases of the standard Sensory Organization Test, with eyes closed for events, with the task of shaking the head.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boyd-Clark LC, Briggs CA, Galea MP. Muscle spindle distribution, morphology, and density in longus colli and multifidus muscles of the cervical spine. Spine (Phila Pa 1976). 2002 Apr 1;27(7):694-701. doi: 10.1097/00007632-200204010-00005. PMID 11923661
- [Result] Peterson BW, Goldberg J, Bilotto G, Fuller JH. Cervicocollic reflex: its dynamic properties and interaction with vestibular reflexes. J Neurophysiol. 1985 Jul;54(1):90-109. doi: 10.1152/jn.1985.54.1.90. PMID 3162006
- [Result] Jull GA, Richardson CA. Motor control problems in patients with spinal pain: a new direction for therapeutic exercise. J Manipulative Physiol Ther. 2000 Feb;23(2):115-7. PMID 10714539
- [Result] Panjabi MM. The stabilizing system of the spine. Part I. Function, dysfunction, adaptation, and enhancement. J Spinal Disord. 1992 Dec;5(4):383-9; discussion 397. doi: 10.1097/00002517-199212000-00001. PMID 1490034
- [Result] Adams M. Re: Spine stability: the six blind men and the elephant. Clin Biomech (Bristol). 2007 May;22(4):486; author reply 487-8. doi: 10.1016/j.clinbiomech.2007.01.001. Epub 2007 Feb 16. No abstract available. PMID 17306912
- [Result] Beinert K, Keller M, Taube W. Neck muscle vibration can improve sensorimotor function in patients with neck pain. Spine J. 2015 Mar 1;15(3):514-21. doi: 10.1016/j.spinee.2014.10.013. Epub 2014 Oct 22. PMID 25452010
- [Result] Brumagne S, Cordo P, Lysens R, Verschueren S, Swinnen S. The role of paraspinal muscle spindles in lumbosacral position sense in individuals with and without low back pain. Spine (Phila Pa 1976). 2000 Apr 15;25(8):989-94. doi: 10.1097/00007632-200004150-00015. PMID 10767813
- [Result] Bosco C, Colli R, Introini E, Cardinale M, Tsarpela O, Madella A, Tihanyi J, Viru A. Adaptive responses of human skeletal muscle to vibration exposure. Clin Physiol. 1999 Mar;19(2):183-7. doi: 10.1046/j.1365-2281.1999.00155.x. PMID 10200901
- [Result] Cardinale M, Bosco C. The use of vibration as an exercise intervention. Exerc Sport Sci Rev. 2003 Jan;31(1):3-7. doi: 10.1097/00003677-200301000-00002. PMID 12562163
- [Result] Torvinen S, Kannus P, Sievanen H, Jarvinen TA, Pasanen M, Kontulainen S, Jarvinen TL, Jarvinen M, Oja P, Vuori I. Effect of four-month vertical whole body vibration on performance and balance. Med Sci Sports Exerc. 2002 Sep;34(9):1523-8. doi: 10.1097/00005768-200209000-00020. PMID 12218749
- [Result] Bruyere O, Wuidart MA, Di Palma E, Gourlay M, Ethgen O, Richy F, Reginster JY. Controlled whole body vibration to decrease fall risk and improve health-related quality of life of nursing home residents. Arch Phys Med Rehabil. 2005 Feb;86(2):303-7. doi: 10.1016/j.apmr.2004.05.019. PMID 15706558
- [Result] Cheng CF, Cheng KH, Lee YM, Huang HW, Kuo YH, Lee HJ. Improvement in running economy after 8 weeks of whole-body vibration training. J Strength Cond Res. 2012 Dec;26(12):3349-57. doi: 10.1519/JSC.0b013e31824e0eb1. PMID 22344045
- [Result] Yong MS, Lee HY, Ryu YU, Lee MY. Effects of craniocervical flexion exercise on upper-limb postural stability during a goal-directed pointing task. J Phys Ther Sci. 2015 Jun;27(6):2005-7. doi: 10.1589/jpts.27.2005. Epub 2015 Jun 30. PMID 26180368
- [Result] Wrisley DM, Stephens MJ, Mosley S, Wojnowski A, Duffy J, Burkard R. Learning effects of repetitive administrations of the sensory organization test in healthy young adults. Arch Phys Med Rehabil. 2007 Aug;88(8):1049-54. doi: 10.1016/j.apmr.2007.05.003. PMID 17678669